CLINICAL TRIAL: NCT05589038
Title: A Randomized, Evaluator-Blinded, Clinical Evaluation of a Regimen of a Baby Wash/Shampoo and Baby Lotion Versus Baby Wash/Shampoo Alone for Tolerability and Impact on Skin Barrier and Microbiome on Newborns
Brief Title: A Study of a Baby Wash/Shampoo and Baby Lotion Versus Baby Wash/Shampoo Alone for Impact on Skin Barrier and Microbiome on Newborns
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to project timelines.
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CCSSKB005013; CCSSKB005013 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2022-10-14; First posted 2022-10-21 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baby Wash/Shampoo (Experimental): Parent participant will bathe the baby participants using baby wash/shampoo at least 3 times per week, but no more than once daily, up to 4 weeks.
  Interventions: Other: Baby Wash/Shampoo
- Baby Wash/Shampoo + Baby Lotion (Experimental): Parent participant will bathe the baby participants using baby wash/shampoo at least 3 times per week, but no more than once daily, and apply lotion at least once daily after bathing, for 4 weeks.
  Interventions: Other: Baby Wash/Shampoo; Other: Baby Lotion

INTERVENTIONS:
Other: Baby Wash/Shampoo — Parent participant will bathe the baby participant with the baby wash/shampoo at least 3 times per week, but no more than once daily.
Other: Baby Lotion — Parent participant will use the baby lotion on baby participants at least once daily.
  Arms: Baby Wash/Shampoo + Baby Lotion

SUMMARY:
The purpose of this study is to demonstrate the tolerance of a baby wash/shampoo alone and the tolerance of a regimen of a baby wash/shampoo and baby lotion in a newborn population.

ELIGIBILITY:
Inclusion Criteria:

For Baby and Parent:

* Baby medically determined to be in overall good health and eligible for study participation. Parent determined to be in generally good health and able to participate fully in the study

For Baby only:

* Healthy, full-term, newborns 0 - 28 days old at start of study, (both vaginal and Caesarean mode of delivery may be included, 37+ weeks gestation)
* Fitzpatrick Skin Types I - VI

For Parent only:

* 18 years of age or older
* Biological, legal guardian and primary caregiver of the baby participant (must be able to present proof of guardianship [that is, birth certificate along with valid identification {ID} of parent, hospital records, insurance card, et cetera {etc.}])
* Able to read, write, speak, and understand english
* Has signed the informed consent document (ICD) including Health Insurance Portability and Accountability Act (HIPAA) disclosure
* Has to have access to internet to be able to complete questionnaires and diaries
* Intends to successfully complete the study and is willing and able to follow the participant responsibilities

Exclusion Criteria:

For Baby and Parent:

* Has known allergies or adverse reactions to common topical skincare products or ingredients in the investigational study materials
* Has self-reported Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication
* Is taking medications that would mask an adverse event (AE) or influence the study results, including: immunosuppressive and steroidal drugs within 3 months before Visit 1 and during the study; non-steroidal anti-inflammatory drugs within 5 days before Visit 1 and during the study; antihistamines within 2 weeks before Visit 1 and during the study; systemic or topical over-the-counter (OTC) or prescription medications that, in the principle investigator (PI)'s judgement, will affect skin condition or interfere with study evaluation (example, antibiotics). Use of acetaminophen as needed is acceptable if it was instructed by the baby's pediatrician. Child vitamins are allowed
* Has a history of or a concurrent health condition/situation which, in the opinion of the PI, may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study
* Is simultaneously participating in any other type of study or has participated in a study within the past 14 days
* Is an employee/contractor or immediate family member of the PI, study site or sponsor

For Baby only:

* Presents with a skin condition that may influence the outcome of the study (example, psoriasis, eczema, atopic dermatitis, cutaneous xerosis, erythema, or active skin cancer)
* Either biological parent or a sibling has clinically determined atopic dermatitis or asthma
* Clinical grade greater than 0 for rash/irritation or greater or equal to 1 for any of the other clinically assessed parameters

For Parent only:

* Is self-reported to be pregnant or planning to become pregnant during the study

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Clinical Assessment of Cutaneous Tolerance scores | Baseline (Day 0) up to Day 28
  The investigator will assess baby's scalp, face, arms, legs, and torso (chest and back) globally for the following parameters (that is, dryness, redness/erythema, rash/irritation, and tactile roughness) on a 4-point scale from '0' (none) to '3' (severe). A decrease in scores indicates an improvement.
Change from Baseline in Parental Assessment Score | Baseline (Day 0) up to Day 28
  The parental assessment for the baby's skin will be performed for burning/stinging and itching on the scalp, face, arms, legs, and torso (chest and back together) on a 4-point scale of '0' (none) to '3' (severe). A decrease in scores indicates an improvement.

SECONDARY OUTCOMES:
Change from Baseline in Microbiome | Baseline (Day 0) up to Day 28
  Change in microbiome samples as analyzed in laboratory will be reported.
Change from Baseline in Metabolome | Baseline (Day 0) up to Day 28
  Change in metabolome samples as analyzed in laboratory will be reported.
Change from Baseline in Skin pH | Baseline (Day 0) up to Day 28
  Change from baseline in skin pH will be reported.
Change from Baseline in Parentype Questionnaire | Baseline (Day 0) up to Day 28
  Parentype questionnaire will be completed by the participant's parent. The six axes will be calculated based on parent's responses on well-being, adaptiveness, parental identity, resilience, sense of ease and parental confidence in intuition and the average will be reported.
Weekly Diary Compliance | Day 1 through Day 28
  The parent participants will be contacted by the site via a phone call visit to complete a weekly diary. Weekly diary compliance will be assessed as follows: Usage compliance for 1 week will include 3 times usage for the Baby Wash/Shampoo and 7 time usage for the Baby Lotion per week. 90 percent (%) compliance would be about 2 time usage misses for the baby wash/shampoo in 28 days, and 3 time usage misses for the Baby lotion.
Product Questionnaire as Assessed by Parent Participants | Day 28
  Product questionnaire will be completed by the parent participants which include the question about "how much do you agree or disagree after using the baby wash/shampoo and baby lotion routine" where 1 indicates "strongly disagree", 2 indicates "somewhat disagree", 3 indicates "neither agree/disagree, 4 indicates "somewhat agree", and 5 indicate "strongly agree".

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Consumer Inc. (J&JCI) Clinical Trial, Study Director — Johnson & Johnson Consumer Inc. (J&JCI)
Locations (1):
- KGL Skin Study Center, LLC, Newtown Square, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Walters RM, Mao G, Gunn ET, Hornby S. Cleansing formulations that respect skin barrier integrity. Dermatol Res Pract. 2012;2012:495917. doi: 10.1155/2012/495917. Epub 2012 Aug 13. PMID 22927835
- [Background] Telofski LS, Morello AP 3rd, Mack Correa MC, Stamatas GN. The infant skin barrier: can we preserve, protect, and enhance the barrier? Dermatol Res Pract. 2012;2012:198789. doi: 10.1155/2012/198789. Epub 2012 Sep 4. PMID 22988452
- [Background] Capone KA, Friscia DL, Nikolovski J, Telofski LS, Stamatas GN. A randomized clinical study on the effects of emollient use on the developing infant skin microbiome and metabolome. Exp Dermatol. 2023 Jan;32(1):75-77. doi: 10.1111/exd.14684. Epub 2022 Oct 20. No abstract available. PMID 36204776
- [Background] Avi Sadeh, D. Sc., Jodi A. Mindell, Ph.D., and Liat Tikotzky, Ph.D. Brief Infant Sleep Questionnaire - Revised Long Form, version January 2020